CLINICAL TRIAL: NCT04329273
Title: Effects of an 8-week Eccentric and Trunk Stability Exercise Program on Muscle Strength and Postural Stability in U19 Elite Soccer Players
Brief Title: Eccentric and Trunk Stability Exercise Program Effects in Young Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konstantinos Dafkou (Other)
Responsible Party: Sponsor-Investigator, Konstantinos Dafkou, Principal Investigator, Aristotle University Of Thessaloniki
Organization: Aristotle University Of Thessaloniki (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ERC-005/2020
Record Dates: First submitted 2020-03-29; First posted 2020-04-01 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Muscle Strength; Postural Balance
MeSH Terms: interventions — Core Stability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): For the balance exercise the participants will perform one-legged stance of certain duration, on a stable surface.
  For the sliding leg curl exercise the participants lay supine on a mat, wearing only socks in order to create a slippery surface between their heels and the gym floor. The player begins by extending the hip and having the working leg on knee flexion. The contralateral limb is on hip flexion and knee flexion. The base of support is the shoulder blades, the elbows and the heel of the working leg. After assuming this position, the player begins to extend the knee, as slowly as possible, resisting the low friction properties of the ground.
  The core stability program consists of front plank, side planks, supine bridge, leg lowering and superman exercise. These exercises will be performed at the end of the training session, in contrast to the balance and hamstring exercises which will be executed before the training session.
  Interventions: Other: Sliding leg curl; Other: Balance training; Other: Core stability
- Control group (No Intervention): The participants in this group will follow only the usual training program

INTERVENTIONS:
Other: Sliding leg curl — The exercise protocol consists of the following sets and repetitions Week 1- 2 sessions with 2 sets of 6 repetitions Week 2- 2 sessions with 3 sets of 6 repetitions Week 3- 2 sessions with 4 sets of 6 repetitions Week 4- 2 sessions with 4 sets of 8 repetitions Week 5- 2 sessions with 4 sets of 10 repetitions Week 6- 2 sessions with 4 sets of 10 repetitions Week 7- 2 sessions with 4 sets of 8 repetitions Week 8- 2 sessions with 4 sets of 8 repetitions
  Arms: Training group
Other: Balance training — The exercise protocol consists of 2 sessions/week with 4 sets of 30'' single stance.
  Week 1 and 2- 1 set of 30'' single leg stance and 3 sets of 30'' single leg stance and ball kicks with contralateral foot Week 3 and 4- 2 sets of 30'' single leg stance while moving the ball around the leg with the contralateral foot and 2 sets of 30'' single leg stance, moving a ball around the knee with hands and kicking a ball with contralateral foot Week 5 and 6- 2 sets of 30'' single leg stance while giving and receiving hand passes with medicine ball (in couples) and 2 sets of 30'' single leg stance with perturbations (in couples) Week 7 and 8- Same as week 5 and 6 with extra 15" in each repetition
  Arms: Training group
Other: Core stability — The exercise protocol consists of the following sets and repetitions Week 1 and 2- 3 sets of 30'' front plank, 3 sets of 20'' side plank, 2 sets of 30'' superman, 2 sets of 30'' supine bridge and 2 sets of 10 repetitions leg lowering exercise Week 3 and 4- increasing difficulty in 2 of the sets Week 5 and 6- adding 1 more set at each exercise Week 7 and 8- adding 15" in each repetition
  Arms: Training group

SUMMARY:
The purpose of the present study is to investigate the effects of an in-season mixed training program on several physiological parameters of soccer players. Twenty-one U19 elite soccer players recruited and randomly assigned to either an 8-week specific training experimental group or a control group. The program will include an eccentric hamstring exercise, static balance exercises and core muscles strengthening exercises. Isokinetic hamstring and quadriceps strength, single leg static balance and lumbopelvic stability will be measured prior and after the intervention.

DETAILED DESCRIPTION:
A total of 123 male Under-19 (U19) players from several soccer teams were initially invited for participation in the study after signing informed consent forms. following a second contact with the participants, questionnaire forms with inclusion and exclusion criteria were send for completion.

Based on their self-report and a clinical examination by a health professional, of the 103 players, 42 did not meet the inclusion criteria, while 12 players did not participate for personal reasons. Of the remaining 69 players, 48 players were excluded, including 3 players reporting an anterior cruciate ligament reconstruction, 14 because of lower extremity injury led to more than two weeks absence from training and 10 players because of secondary injuries or health problems that led to loss of training the past 3 months.

A neutral, blinded investigator with no further involvement in the study was responsible for randomized allocation of participants in two groups. All training sessions in the training group will be supervised by a fitness coach, who will ensure that the exercises are performed according to protocol.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 19 years old soccer players
* Trained at least 3 times and played 1 match weekly, the past 4 years
* Healthy
* Free from muscle injuries in the 6 months prior to the study

Exclusion Criteria:

* History of anterior cruciate ligament rupture
* History of ankle, hip or knee injury with duration at least 1 week, in the 3 months prior to the study
* Muscle injury with duration at least 1 week, in the 3 months prior to the study
* Any reason resulting in 2 weeks loss of training the preceding 6 months
* Involvement in hamstring strengthening, core stability or balance training program in the 6 months prior to the study

Ages: 16 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-05 (Actual)

PRIMARY OUTCOMES:
Peak concentric and eccentric torque of hamstrings and quadriceps | Change from baseline assessment at 8 weeks
  Peak torque (N.m) is measured using isokinetic dynamometer at each angular velocity (30°·s-1, 180°·s-1, 240°·s-1).
Total sway of the center of pressure (CoP) | Change from baseline assessment at 8 weeks
  This is defined as the average distance (mm) of the CoP from the reference lines and the amplitude is its standard deviation

SECONDARY OUTCOMES:
Angle at peak torque of hamstrings and quadriceps | Change from baseline assessment at 8 weeks
  The angle at which peak torque of hamstrings and quadriceps muscles was achieved, at each angular velocity, measured in degrees (°)
Conventional hamstrings to quadriceps ratio | Change from baseline assessment at 8 weeks
  This is calculated by dividing peak isokinetic concentric hamstring strength by the peak isokinetic concentric quadriceps strength, at the same angular velocity
Dynamic hamstrings to quadriceps ratio | Change from baseline assessment at 8 weeks
  This is calculated by dividing peak isokinetic eccentric hamstring strength by the peak isokinetic concentric quadriceps strength, at the same angular velocity
Mixed hamstrings to quadriceps ratio | Change from baseline assessment at 8 weeks
  This is calculated by dividing peak isokinetic eccentric hamstring strength at 30°·s-1 by the peak isokinetic concentric quadriceps strength at 240°·s-1
Average speed of CoP | Change from baseline assessment at 8 weeks
  This reflects the amplitude and frequency of CoP movements and is calculated as the total length of the path of CoP divided by the test trial time (mm·s-1 )

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Dafkou, Principal Investigator — Laboratory of Neuromechanics, Aristotle University of Thessaloniki
Locations (1):
- Laboratory of Neuromechanics, Department of physical education and sport sciences, Aristotle University of Thessaloniki, Serres, Greece

IPD SHARING:
Plan to Share IPD: No